CLINICAL TRIAL: NCT03591822
Title: Prevention of Care-induced Pain in Elderly Persons With Cognitive Impairments and Living in EHPAD : Systematic Evaluation and Mediation With the PARO Robot.
Brief Title: Pilot Study of a Robot-assisted Intervention for the Management of Care-induced Pain in Dementia
Acronym: PARODOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: The Paul Bennetot Foundation (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: K170608J
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Moderate to Severe Dementia
Keywords: Dementia; Pain; Nursing care; Psychosocial intervention; Robot-assisted therapy; paro robot
MeSH Terms: conditions — Dementia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm AB : Intervention under study x Control intervention (Other): Subjects receive intervention A during which they will benefit from a systemic pain assessment and from the PARO robot as a therapeutic mediator, followed by intervention B during which patients will benefit from a systemic pain assessment without the PARO robot.
  Interventions: Behavioral: A : Systemic evaluation of the pain and mediation with the PARO therapeutic robot; Behavioral: B : Systemic evaluation of the pain
- Arm BA: Control intervention x Intervention under study (Other): Subjects receive intervention B during which they will benefit from a systemic pain assessment without the PARO robot, followed by intervention A during which patients will benefit from a systemic pain assessment and from the PARO robot as a therapeutic mediator.
  Interventions: Behavioral: A : Systemic evaluation of the pain and mediation with the PARO therapeutic robot; Behavioral: B : Systemic evaluation of the pain

INTERVENTIONS:
Behavioral: A : Systemic evaluation of the pain and mediation with the PARO therapeutic robot — Each session with the PARO robot will encompasses the same four following steps (a) Meeting Paro (b) Proposing contact (c) Individually using Paro during the care (d) End of the exposure.
Behavioral: B : Systemic evaluation of the pain — A systematic evaluation of the pain

SUMMARY:
Health care professionals lack tools to deal with acute pain in patients with moderate to severe dementia during daily nursing situations. Care-induced pain in institutionalized persons with cognitive impairments can cause anxiety and behavioral problems.The aim of this study is to demonstrate that a systematic identification of pain associated with the use of social robots such as the PARO robot may contribute to a better anticipation and management of care-induced pain. The investigators hypothesize that an individual use of the PARO robot would bring relaxation to the patient, a distraction regarding the aversive situation of care and, thus, it would prevent manifestations of acute pain in patients with dementia.

Secondary objectives of the study :

1. determine the effect of the use of PARO during painful cares on quality of life, medication of patients, and perceived workload of the health-care team.
2. examine socio-demographic and clinical responders' participants to the intervention, and,
3. identify essential elements regarding cost-effectiveness of a systematic evaluation of pain and a mediation with the PARO robot in care-induced pain

DETAILED DESCRIPTION:
in is a frequent problem in persons with moderate to severe dementia and has been associated to different care situations. Daily observations in care homes show that pain frequently causes anxiety and behavioral symptoms, including agitation and opposition to nursing care. A key recommendation of the International Psychogeriatric Association (IPA) is the use of psychosocial approaches as first-line therapy for behavioral problems in persons with dementia. Indeed, a wide range of non-pharmacological interventions for persons with dementia exist, such as biofeedback, music therapy, therapeutic touch or relaxation. Most of these interventions have shown positive results on health status, quality of life, socialization, and functional capacity in dementia. However, to date, little is known on the effect of psychosocial interventions on care-induced pain in this population. In consequence, there is still a need for the development of innovative interventions.

At a time when modern technologies are assuming a central role in our society, investigators are currently witnessing an important evolution of the use of social robots in healthcare interventions. In this research area, numerous studies have been conducted with social robots, such as PARO®, an animal-like robot modeled on a baby harp seal. Most of them have been successful in encouraging communication and/or social behaviors and also reducing Behavioral and Psychological Symptoms of Dementia (BPSD), loneliness, stress' levels, agitation and the use of pain medication. However, although these results indicate a potential application of robot-assisted therapies for pain management in persons with dementia, the use of PARO during painful care-situations is still to be investigated.

The investigators propose a new combination of current health cares, namely to mediate care-induced pain with the PARO robot.

Consequently, a randomized AB/BA crossover design will be employed. Patients will be assigned randomly to either phase A during which they will benefit from a systemic pain assessment and from the PARO robot as a therapeutic mediator, followed by phase B during which patients will benefit from a systemic pain assessment without the PARO robot, or phase B followed by phase A.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 60 years of age
* Consent to participate
* Patient diagnosed by a geriatrician or a neurologist with moderate to severe dementia (MMSE<24), according to the criteria of the Diagnostic and Statistical Manual DSM IV-TR (APA,2004) and NINCDS-ADRDA(McKhann et al.1984).
* Patient living in a nursing home or a long stay department
* Painful patient during nursing care (pain drugs prescription or direct observation)

Exclusion Criteria:

* Patient (or patient's legal representative) does not provide consent
* The presence of acute organic disease or psychiatric decompensation and major neuropsychiatric symptoms incompatible with the intervention.
* Patient who cannot interact physically with Paro
* The presence of multidrug-resistant bacteria in patient to reduce the risk of contamination.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
ALGOPLUS scale | 2 months
  A proximal measure of pain rating on a scale of 1) facial expressions, 2) look, 3) complaints, 4) body position and, 5) atypical behaviors.
  And a distal measures of pain

SECONDARY OUTCOMES:
PACSLAC-F score | at inclusion
  A distal measure of pain .
PACSLAC-F score | 4 weeks
  A distal measure of pain .
PACSLAC-F score | 8 weeks
  A distal measure of pain .
Simple verbal scale (SVS) | 2 months
  Measurement with a scale in 3 points
The appreciation of the Paro robot | 2 months
  Measurement with a visual scale in 5 points: from 1 (not at all) to 5 (considerably) on a visual scale.
Incidence of patient Medication | 2 months
  Medications (analgesic, neuroleptic, anxiolytic, antidepressant, sleeping pill) taken by the patient
EQ-5D score | at inclusion
  A questionnaire (EQ-5D) of quality life which includes five single-item dimensions assessing: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression of participants.
EQ-5D score | 4 weeks
  A questionnaire (EQ-5D) of quality life which includes five single-item dimensions assessing: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression of participants.
EQ-5D score | 8 weeks
  A questionnaire (EQ-5D) of quality life which includes five single-item dimensions assessing: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression of participants.
Appreciation of care | 2 months
  Measurement with 2 visual scales in 4 and 5 points
Appreciation of PARO robot | 2 months
  Measurement with a visual scale in 5 points
Duration of the care | 2 months
NASA-TLX score | 2 months
  The NASA-TLX is an instrument to assess overall subjective workload with 6 dimensions of "workload" experienced by the health-care team: Mental Demand, Physical Demand and Temporal Demand, Frustration, Effort, and Performance

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie RIGAUD, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (5):
- France (5):
  - Résidence Mutualiste " L'adret ", Bellegarde-en-Forez
  - Résidence Mutualiste " Les Tilleuls ", La Grand-Croix
  - Hôpital Broca, Paris
  - Résidence Mutualiste " La Cerisaie ", Saint-Etienne
  - Résidence Mutualiste " Marie Lagrevol ", Saint-Just-Malmont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Demange M, Pino M, Kerherve H, Rigaud AS, Cantegreil-Kallen I. Management of acute pain in dementia: a feasibility study of a robot-assisted intervention. J Pain Res. 2019 Jun 7;12:1833-1846. doi: 10.2147/JPR.S179640. eCollection 2019. PMID 31289446